CLINICAL TRIAL: NCT04047472
Title: A Twelve-Month, Randomized, Double-Masked, Multicenter, Phase III, Two-Arm Study Comparing the Efficacy and Safety of Brolucizumab 6 mg Versus Aflibercept in Chinese Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Study of Efficacy and Safety of Brolucizumab vs. Aflibercept in Chinese Patients With Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRTH258A2307
Record Dates: First submitted 2019-07-01; First posted 2019-08-06 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Macular degeneration; age-related macular degeneration (AMD); vision loss; macula damage; retina damage; wet macular degeneration; AMD
MeSH Terms: conditions — Macular Degeneration; Vision Disorders; Wet Macular Degeneration | interventions — brolucizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg (Experimental): 3 monthly intravitreal injections of brolucizumab 6 mg in the loading treatment period (q4w regimen) up to Week 8 followed by injections every 12 weeks (q12w regimen) or 8 weeks (q8w) up to Week 40 or Week 44, depending on disease activity status.
  Interventions: Drug: Brolucizumab 6mg
- Aflibercept 2 mg (Active Comparator): 3 monthly intravitreal injections of aflibercept 2 mg in the loading treatment period (q4w regimen) up to Week 8 followed by injections every 8 weeks (q8w) up to Week 40.
  Interventions: Drug: Aflibercept 2 mg

INTERVENTIONS:
Drug: Brolucizumab 6mg — Intravitreal injection
  Other Names: Beovu
  Arms: Brolucizumab 6 mg
Drug: Aflibercept 2 mg — Intravitreal injection
  Other Names: Eylea
  Arms: Aflibercept 2 mg

SUMMARY:
To compare brolucizumab to aflibercept in Chinese patients with untreated active choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD)

DETAILED DESCRIPTION:
This was a randomized, double-masked, multicenter, parallel-group, active-controlled study. The study included 14 scheduled visits over 48 weeks. After confirmation of eligibility at baseline, participants were randomized in a 1:1 ratio to one of the 2 treatment arms:

* Brolucizumab 6 mg: 3 monthly intravitreal injections of brolucizumab 6 mg in the loading treatment period (q4w regimen) up to Week 8 followed by injections every 12 weeks (q12w regimen) or 8 weeks (q8w) up to Week 40 or Week 44, depending on disease activity status.
* Aflibercept 2 mg: 3 monthly intravitreal injections of aflibercept 2 mg in the loading treatment period (q4w regimen) up to Week 8 followed by injections every 8 weeks (q8w) up to Week 40. Disease activity assessments (DAAs) were conducted by the masked investigator for both treatment arms at Weeks 16, 20, 32 and 44 to determine the regimen of brolucizumab arm (i.e., q12w or q8w).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment was performed.
* Male or female Chinese participants ≥ 50 years of age at the time of screening.
* Active CNV lesions secondary to AMD that affect the central subfield (including retinal angiomatous proliferation lesions with a CNV component) in the study eye at screening and confirmed by the Central Reading Center (CRC).
* Total area of CNV (including both classic and occult components) must comprise > 50% of the total lesion area in the study eye at screening and confirmed by the CRC.
* Intra and/or subretinal fluid affecting the central subfield of the study eye at screening and confirmed by the CRC.
* BCVA between 78 and 23 letters, inclusive, in the study eye at screening and baseline using ETDRS testing.

Exclusion Criteria:

* Any active intraocular or periocular infection or active intraocular inflammation (e.g., infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in study eye at baseline.
* Central subfield of the study eye affected by fibrosis or geographic atrophy assessed by color fundus photography at screening and confirmed by the CRC.
* Total area of fibrosis ≥ 50% of the total lesion in the study eye at screening and confirmed by the CRC.
* Subretinal blood affecting the foveal center point and/or ≥ 50% of the lesion of the study eye at screening and confirmed by the CRC.
* Previous treatment with any approved or investigational drugs for nAMD in the study eye (other than vitamin supplements).
* Retinal pigment epithelium rip/tear in the study eye at screening.
* Current vitreous hemorrhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to baseline.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- China (19):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Yixing, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xi'an, Shaanxi
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://clinicalstudydatarequest.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Started | 199 | 198
Completed | 183 | 182
Not Completed | 16 | 16
Not completed — Adverse Event | 3 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg | Total
Number analyzed (Participants) | 199 | 198 | 397
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.1 (7.58) | 68.0 (7.68) | 68.5 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 54 | 124
  Male | 129 | 144 | 273
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 199 | 198 | 397
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 48 in Best-Corrected Visual Acuity in Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score between 78 and 23 ETDRS letters (inclusive) at Screening and Baseline in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better functioning.
  Last observation carried forward (LOCF) was used for the imputation of missing values.
Time Frame: Baseline, Week 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Letters Read
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Letters Read | 9.9 (0.82) | 10.9 (0.82)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — Non-inferiority of brolucizumab to aflibercept with respect to change from baseline in BCVA, considering a margin of 4 letters; p = 0.006, ANOVA; LS mean difference = -1.1, 90% CI 2-sided [-3.0 to 0.9], Standard Error of Mean 1.16

2. Secondary Outcome: Average Change From Baseline Over the Period of Week 36 to Week 48 in Best-Corrected Visual Acuity in Study Eye
Description: as for outcome 1
Time Frame: Baseline, over the period Week 36 to Week 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Letters Read
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Letters Read | 9.7 (0.78) | 11.0 (0.79)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.009, ANOVA; LS mean difference = -1.4, 90% CI 2-sided [-3.2 to 0.5], Standard Error of Mean 1.11

3. Secondary Outcome: q12w Treatment Status at Week 48 (for Subjects Randomized to Brolucizumab 6 mg Only) - Probability
Description: The estimate for the proportion of participants with a positive q12w treatment status was derived from Kaplan-Meier time-to-event analyses for the event "first q8w-need", applying a "q8w-need" allocation in case of missing or confounded data attributable to lack of efficacy and/or lack of safety for the purpose of analysis. The proportion of participants with a positive q12w treatment status was derived as follows according to the "sufficient efficacy and safety" approach: the q8w-need assessment was imputed as "Yes" at the disease activity assessment (DAA) visit following early treatment/study discontinuation due to lack of efficacy and /or lack of safety of the study treatment (applicable to both missing and non-missing DAAs).
Time Frame: Week 44
Population: Full Analysis Set (FAS)
Measure: Number (90% Confidence Interval); unit: Probability of no q8w-need
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 199
Probability of no q8w-need | 0.595 [0.529 to 0.655]

4. Secondary Outcome: q12w Treatment Status at Week 48 Within the Subjects With no q8w Need During the First q12w Cycle (Week 16 and Week 20) (for Subjects Randomized to Brolucizumab 6 mg Only) - Probability
Description: The estimate for the proportion of participants with a positive q12w treatment status was derived from Kaplan-Meier time-to-event analyses for the event "first q8w-need", applying a "q8w-need" allocation in case of missing or confounded data attributable to lack of efficacy and/or lack of safety for the purpose of analysis.
  The analysis of "q12w treatment status within the participants randomized to brolucizumab 6 mg and with no q8w need during the first q12w cycle" was based on the subset of FAS participants randomized to brolucizumab 6 mg with no identified q8w-need at Week 16 and Week 20.
Time Frame: Week 44
Population: FAS - Participants in the FAS randomized to brolucizumab 6 mg with no identified q8w-need at Week 16 and Week 20.
Measure: Number (90% Confidence Interval); unit: Probability of no q8w-need
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 117
Probability of no q8w-need | 0.860 [0.791 to 0.908]

5. Secondary Outcome: Number (%) of Participants With q8w Treatment Need as Assessed by the Investigator at First Disease Activity Assessment (DAA) Visit
Description: For both arms, the treatment was initiated with 3 monthly injections at Weeks 0, 4 and 8 (loading phase). Week 12 was scheduled as a "no injection visit" for both arms per protocol. Therefore, by Week 16, the planned treatment exposure was identical between the treatment arms, allowing a matched comparison of brolucizumab and aflibercept up to 8 weeks after loading.
Time Frame: Week 16
Population: Full Analysis Set (FAS) - for participants with a valid measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 181 | 185
Participants | 30 | 47

6. Secondary Outcome: Change From Baseline at Each Study Visit in Best-Corrected Visual Acuity in Study Eye
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Letters Read
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Letters Read
  Week 4 | 3.9 (0.58) | 4.2 (0.58)
  Week 8 | 6.1 (0.61) | 6.5 (0.61)
  Week 12 | 7.4 (0.69) | 8.4 (0.69)
  Week 16 | 8.3 (0.74) | 9.4 (0.74)
  Week 20 | 8.2 (0.78) | 10.5 (0.79)
  Week 24 | 8.3 (0.81) | 10.0 (0.81)
  Week 28 | 9.1 (0.77) | 11.0 (0.77)
  Week 32 | 9.2 (0.78) | 10.7 (0.78)
  Week 36 | 9.1 (0.79) | 11.1 (0.80)
  Week 40 | 9.7 (0.79) | 10.9 (0.79)
  Week 44 | 10.0 (0.80) | 11.2 (0.80)

7. Secondary Outcome: Average Change From Baseline in Best Corrected Visual Acuity (Letters Read) From Week 4 or Week 12 up to Week 48 for the Study Eye
Description: as for outcome 1
Time Frame: Baseline, over the period of Week 4 or Week 12 to Week 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Letters Read
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Letters Read
  Average change from baseline over the period Week 4 through Week 48 | 8.3 (0.68) | 9.6 (0.68)
  Average change from baseline over the period Week 12 through Week 48 | 8.9 (0.73) | 10.4 (0.74)

8. Secondary Outcome: Number of Subjects With Best-Corrected Visual Acuity of 73 Letters or More at Each Visit
Description: as for outcome 1
Time Frame: Baseline up to Week 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Week 4 | 36 | 50
  Week 8 | 47 | 60
  Week 12 | 59 | 70
  Week 16 | 69 | 74
  Week 20 | 68 | 86
  Week 24 | 68 | 78
  Week 28 | 73 | 82
  Week 32 | 73 | 85
  Week 36 | 71 | 87
  Week 40 | 73 | 84
  Week 44 | 78 | 92
  Week 48 | 72 | 86

9. Secondary Outcome: Gain in BCVA (Letters Read): Number (%) of Participants Who Gained ≥ 5, ≥ 10 and ≥ 15 Letters in Best-correct Visual Acuity From Baseline or Reached BCVA ≥ 84 Letters at Week 48 for the Study Eye
Description: as for outcome 1
Time Frame: Baseline up to Week 48
Population: Full Analysis Set (FAS) Last Observation carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Participants with ≥ 5 letters gain from baseline or reached BCVA of ≥ 84 letters at Week 48 | 139 | 146
  Participants with ≥ 10 letters gain from baseline or reached BCVA of ≥ 84 letters at Week 48 | 103 | 104
  Participants with ≥ 15 letters gain from baseline or reached BCVA of ≥ 84 letters at Week 48 | 68 | 73

10. Secondary Outcome: Gain in BCVA (Letters Read): Number (%) of Participants Who Gained ≥ 5 Letters in Best-correct Visual Acuity From Baseline or Reached BCVA >=84 Letters at the Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Week 4 | 73 | 94
  Week 8 | 102 | 115
  Week 12 | 122 | 139
  Week 16 | 134 | 149
  Week 20 | 133 | 147
  Week 24 | 129 | 149
  Week 28 | 134 | 147
  Week 32 | 131 | 154
  Week 36 | 129 | 151
  Week 40 | 134 | 152
  Week 44 | 136 | 151
  Week 48 | 139 | 146

11. Secondary Outcome: Gain in BCVA (Letters Read): Number (%) of Participants Who Gained ≥ 10 Letters in Best-correct Visual Acuity From Baseline or Reached BCVA >=84 Letters at the Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Week 4 | 39 | 35
  Week 8 | 57 | 59
  Week 12 | 79 | 85
  Week 16 | 88 | 93
  Week 20 | 86 | 107
  Week 24 | 90 | 98
  Week 28 | 91 | 108
  Week 32 | 95 | 107
  Week 36 | 94 | 108
  Week 40 | 102 | 98
  Week 44 | 101 | 107
  Week 48 | 103 | 104

12. Secondary Outcome: Gain in BCVA (Letters Read): Number (%) of Participants Who Gained ≥ 15 Letters in Best-correct Visual Acuity From Baseline or Reached BCVA >=84 Letters at the Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Week 4 | 21 | 19
  Week 8 | 37 | 28
  Week 12 | 49 | 48
  Week 16 | 56 | 55
  Week 20 | 57 | 59
  Week 24 | 57 | 54
  Week 28 | 61 | 64
  Week 32 | 62 | 64
  Week 36 | 64 | 69
  Week 40 | 66 | 68
  Week 44 | 63 | 69
  Week 48 | 68 | 73

13. Secondary Outcome: Loss in BCVA (Letters Read): Number (%) of Participants Who Lost ≥ 5, ≥ 10 and ≥ 15 Letters in Best-correct Visual Acuity From Baseline at Week 48 for the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Week 48
Population: Full Analysis Set (FAS) Last Observation carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Participants with ≥ 5 letters loss from baseline at Week 48 | 16 | 11
  Participants with ≥ 10 letters loss from baseline at Week 48 | 7 | 6
  Participants with ≥ 15 letters loss from baseline at Week 48 | 5 | 4

14. Secondary Outcome: Loss in BCVA (Letters Read): Number (%) of Participants Who Lost ≥ 5 Letters in Best-correct Visual Acuity From Baseline to Each Post-baseline Visit for the Study
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Week 4 | 20 | 15
  Week 8 | 19 | 15
  Week 12 | 14 | 8
  Week 16 | 18 | 10
  Week 20 | 20 | 8
  Week 24 | 18 | 13
  Week 28 | 17 | 9
  Week 32 | 14 | 13
  Week 36 | 15 | 10
  Week 40 | 13 | 10
  Week 44 | 14 | 9
  Week 48 | 16 | 11

15. Secondary Outcome: Loss in BCVA (Letters Read): Number (%) of Participants Who Lost ≥ 10 Letters in Best-correct Visual Acuity From Baseline to Each Post-baseline Visit for the Study
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Week 4 | 6 | 6
  Week 8 | 5 | 4
  Week 12 | 6 | 4
  Week 16 | 6 | 4
  Week 20 | 9 | 5
  Week 24 | 13 | 5
  Week 28 | 8 | 4
  Week 32 | 9 | 5
  Week 36 | 8 | 5
  Week 40 | 6 | 6
  Week 44 | 7 | 6
  Week 48 | 7 | 6

16. Secondary Outcome: Loss in BCVA (Letters Read): Number (%) of Participants Who Lost ≥ 15 Letters in Best-correct Visual Acuity From Baseline to Each Post-baseline Visit for the Study
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Week 4 | 2 | 5
  Week 8 | 2 | 3
  Week 12 | 5 | 3
  Week 16 | 6 | 4
  Week 20 | 7 | 4
  Week 24 | 9 | 3
  Week 28 | 5 | 4
  Week 32 | 5 | 3
  Week 36 | 6 | 2
  Week 40 | 6 | 4
  Week 44 | 5 | 3
  Week 48 | 5 | 4

17. Secondary Outcome: Average Change From Baseline Over the Period Week 4 Through Week 48 in Central Subfield Thickness - Total in Study Eye
Description: Central Subfield Thickness Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
  Central subfield thickness (CSFT) is a key anatomical parameter of central macula and is the average thickness in the center subfield as measured from the Internal Limiting Membrane (ILM) to the Bruch's Membrane (BM). The center subfield is the circular region centered on the anatomic fovea with the radius of 500 μm.
Time Frame: Baseline, over the period Week 4 through Week 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
μm | -181.2 (7.46) | -161.9 (7.48)

18. Secondary Outcome: Average Change From Baseline Over the Period Week 36 Through 48 in Central Subfield Thickness - Total in Study Eye
Description: as for outcome 17
Time Frame: Baseline, over the period Week 36 to Week 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
μm | -187.9 (8.38) | -167.2 (8.40)

19. Secondary Outcome: Change From Baseline at Each Study Visit in Central Subfield Thickness - Total in Study Eye
Description: as for outcome 17
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
μm
  Week 4 | -148.5 (6.50) | -132.5 (6.51)
  Week 8 | -183.3 (6.95) | -161.8 (6.97)
  Week 12 | -193.2 (7.22) | -169.9 (7.24)
  Week 16 | -179.5 (7.99) | -152.6 (8.01)
  Week 20 | -172.2 (7.91) | -175.6 (7.93)
  Week 24 | -185.2 (8.33) | -152.0 (8.35)
  Week 28 | -186.8 (8.06) | -172.0 (8.08)
  Week 32 | -174.0 (8.37) | -157.2 (8.39)
  Week 36 | -191.2 (8.29) | -171.3 (8.31)
  Week 40 | -184.6 (8.57) | -159.0 (8.59)
  Week 44 | -184.7 (8.64) | -175.3 (8.66)
  Week 48 | -191.1 (8.71) | -163.2 (8.73)

20. Secondary Outcome: Change From Baseline at Each Study Visit in Central Subfield Thickness - Neurosensory Retina (μm) in Study Eye
Description: Central Subfield Thickness Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
  The central subfield thickness-neurosensory retina (CSFTns) is the average thickness in the center subfield as measured from the Internal Limiting Membrane (ILM) to the outer segment tips.
  The center subfield is the circular region centered on the anatomic fovea with the radius of 500μm.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
μm
  Week 4 | -57.2 (4.55) | -48.3 (4.57)
  Week 8 | -65.4 (4.94) | -53.2 (4.95)
  Week 12 | -68.6 (5.11) | -53.2 (5.12)
  Week 16 | -63.8 (5.22) | -48.4 (5.24)
  Week 20 | -60.8 (5.44) | -56.4 (5.45)
  Week 24 | -67.0 (5.22) | -49.9 (5.23)
  Week 28 | -67.2 (5.28) | -54.5 (5.29)
  Week 32 | -62.7 (5.26) | -50.1 (5.27)
  Week 36 | -69.2 (5.42) | -56.3 (5.43)
  Week 40 | -67.9 (5.45) | -52.7 (5.46)
  Week 44 | -67.8 (5.53) | -57.2 (5.54)
  Week 48 | -69.7 (5.38) | -53.0 (5.39)

21. Secondary Outcome: Number of Participants With Presence of Subretinal Field (SRF) and/or Intraretinal Fluid (Central Subfield) (IRF) in the Study Eye at Each Postbaseline Visit (and Specifically Week 16 and Week 48)
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Week 4 | 78 | 92
  Week 8 | 32 | 51
  Week 12 | 33 | 44
  Week 16 | 41 | 63
  Week 20 | 55 | 37
  Week 24 | 39 | 63
  Week 28 | 44 | 40
  Week 32 | 55 | 57
  Week 36 | 37 | 40
  Week 40 | 40 | 56
  Week 44 | 45 | 37
  Week 48 | 35 | 52

22. Secondary Outcome: Number of Participants With Absence of Subretinal Field (SRF) and Intraretinal Fluid (Central Subfield) (IRF) in the Study Eye Between Week 36 and Week 48
Time Frame: Between Weeks 36 and Weeks 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  0 visits with no fluid between Week 36 to 48 | 18 | 24
  1 visit with no fluid between Week 36 to 48 | 13 | 12
  2 visits with no fluid between Week 36 to 48 | 15 | 18
  3 visits with no fluid between Week 36 to 48 | 16 | 17
  4 visits with no fluid between Week 36 to 48 | 137 | 127

23. Secondary Outcome: Subretinal Fluid (SRF) Status in the Central Subfield: Number of Subjects With Presence of SRF by Visit for the Study Eye
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Baseline | 149 | 156
  Week 4 | 63 | 83
  Week 8 | 19 | 42
  Week 12 | 18 | 34
  Week 16 | 30 | 50
  Week 20 | 35 | 28
  Week 24 | 26 | 49
  Week 28 | 29 | 31
  Week 32 | 34 | 46
  Week 36 | 21 | 35
  Week 40 | 24 | 49
  Week 44 | 27 | 32
  Week 48 | 20 | 43

24. Secondary Outcome: Intraretinal Fluid (IRF) Status in the Central Subfield: Number of Subjects With Presence of IRF by Visit for the Study Eye
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Baseline | 83 | 81
  Week 4 | 26 | 17
  Week 8 | 15 | 13
  Week 12 | 15 | 13
  Week 16 | 13 | 22
  Week 20 | 23 | 10
  Week 24 | 15 | 19
  Week 28 | 15 | 9
  Week 32 | 23 | 14
  Week 36 | 17 | 6
  Week 40 | 21 | 13
  Week 44 | 22 | 7
  Week 48 | 16 | 13

25. Secondary Outcome: Subretinal Pigment Epithelium (Sub-RPE) Fluid Status in the Central Subfield: Number of Subjects With Presence of Sub-RPE by Visit for the Study Eye
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Baseline | 26 | 32
  Week 4 | 11 | 20
  Week 8 | 7 | 17
  Week 12 | 10 | 13
  Week 16 | 12 | 15
  Week 20 | 9 | 9
  Week 24 | 10 | 10
  Week 28 | 6 | 7
  Week 32 | 5 | 10
  Week 36 | 8 | 7
  Week 40 | 6 | 10
  Week 44 | 5 | 8
  Week 48 | 6 | 9

26. Secondary Outcome: Change From Baseline at Weeks 12 and 48 in Choroidal Neovascularization (CNV) Lesion in Study Eye
Time Frame: Baseline, Week 12 and Week 48
Population: Full Analysis Set (FAS) Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
mm^2
  Week 12 | -1.395 (0.1613) | -1.378 (0.1617)
  Week 48 | -2.034 (0.2002) | -1.984 (0.2007)

27. Secondary Outcome: Number of Subjects With Presence of Fibrosis (Central Subfield) in the Study Eye by Visit
Description: As assessed by color fundus photography.
Time Frame: Baseline, Week 12, Week 48
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Baseline | 0 | 0
  Week 12 (n=182, 177): number analyzed (Participants) | 182 | 177
  Week 12 (n=182, 177) | 15 | 17
  Week 48 (n=166,164): number analyzed (Participants) | 166 | 164
  Week 48 (n=166,164) | 18 | 24

28. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Composite Score
Description: The VFQ-25 includes a series of 25 questions pertaining to vision or feelings about a vision condition. Answers are selected among a numbered list of possible responses, the values of which are ultimately recoded and converted to a 0 to 100 scale. Items within each subscale are averaged together to create 12 subscale scores. An overall composite score was calculated by averaging vision-targeted subscale scores, excluding the general health rating question. All items are scored so that a high score represents better visual functioning.
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | 3.0 (13.03) | 3.7 (12.94)
  Week 48 (n=165,159): number analyzed (Participants) | 165 | 159
  Week 48 (n=165,159) | 4.1 (14.00) | 2.9 (13.69)

29. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - General Vision
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | 7.7 (17.88) | 7.8 (17.47)
  Week 48 (n=165,159): number analyzed (Participants) | 165 | 159
  Week 48 (n=165,159) | 9.0 (19.68) | 6.4 (16.89)

30. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Ocular Pain
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | 0.9 (17.68) | 6.1 (15.74)
  Week 48 (n=165,159): number analyzed (Participants) | 165 | 159
  Week 48 (n=165,159) | 1.0 (19.37) | 3.1 (17.88)

31. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Near Activities
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 170 | 167
Scores on a Scale
  Week 24 | 5.3 (22.02) | 5.8 (21.03)
  Week 48 (n=162,157): number analyzed (Participants) | 162 | 157
  Week 48 (n=162,157) | 8.1 (23.28) | 5.7 (22.64)

32. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Distance Activities
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | 2.2 (21.09) | 4.2 (20.07)
  Week 48 (n=163,159): number analyzed (Participants) | 163 | 159
  Week 48 (n=163,159) | 3.8 (20.62) | 4.8 (21.11)

33. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Social Functioning
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | 1.5 (13.44) | 2.4 (14.50)
  Week 48 (n=165,159): number analyzed (Participants) | 165 | 159
  Week 48 (n=165,159) | 2.3 (14.90) | 0.8 (15.83)

34. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Mental Health
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | 4.6 (25.61) | 0.6 (20.34)
  Week 48 (n=165,159): number analyzed (Participants) | 165 | 159
  Week 48 (n=165,159) | 4.7 (22.46) | 1.0 (21.55)

35. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Role Difficulties
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | 0.5 (27.25) | 3.8 (25.91)
  Week 48 (n=165,159): number analyzed (Participants) | 165 | 159
  Week 48 (n=165,159) | 4.5 (25.23) | 2.7 (25.68)

36. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Dependency
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | 3.9 (28.38) | 2.1 (24.29)
  Week 48 (n=165,159): number analyzed (Participants) | 165 | 159
  Week 48 (n=165,159) | 6.6 (27.85) | 0.6 (26.50)

37. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Driving
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 34 | 43
Scores on a Scale
  Week 24 (n=33, 43): number analyzed (Participants) | 33 | 43
  Week 24 (n=33, 43) | 3.4 (15.50) | 0.8 (19.65)
  Week 48 (n=34,37): number analyzed (Participants) | 34 | 37
  Week 48 (n=34,37) | 3.9 (17.28) | 4.6 (15.80)

38. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Color Vision
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 167 | 162
Scores on a Scale
  Week 24 | 1.3 (12.95) | 2.2 (18.36)
  Week 48 (n=161,155): number analyzed (Participants) | 161 | 155
  Week 48 (n=161,155) | 0.6 (15.55) | 0.5 (14.93)

39. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - Peripheral Vision
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 168
Scores on a Scale
  Week 24 | 1.6 (17.76) | 2.4 (16.92)
  Week 48 (n=164,158): number analyzed (Participants) | 164 | 158
  Week 48 (n=164,158) | 0.5 (18.67) | 1.4 (19.60)

40. Secondary Outcome: Change in Subject Reported Outcomes (Visual Function Questionnaire-25) - General Health Rating
Description: as for outcome 28
Time Frame: Baseline, Week 24 and Week 48
Population: Full Analysis Set - Observed - for participants with a valid measurement
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 172 | 169
Scores on a Scale
  Week 24 | -3.6 (24.13) | 0.7 (24.00)
  Week 48 (n=165,159): number analyzed (Participants) | 165 | 159
  Week 48 (n=165,159) | -4.4 (24.84) | -2.7 (26.62)

41. Secondary Outcome: Anti-drug Antibody (ADA): Frequency Distribution of Pre-dose ADA Status in the Brolucizumab Arm
Description: To assess immunogenicity of brolucizumab 6 mg.
Time Frame: Baseline
Population: Safety Analysis Set - for a subset of treated participants with a valid measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 198
Participants
  Pre-dose ADA Status = Negative | 82
  Pre-dose ADA Status = Positive | 116

42. Secondary Outcome: Anti-drug Antibody (ADA): Frequency Distribution of Integrated ADA Status in the Brolucizumab Arm
Description: To assess immunogenicity of brolucizumab 6 mg.
Time Frame: Baseline up to Week 48 (End of Study)
Population: Safety Analysis Set - for a subset of treated participants with a valid measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg
Number analyzed (Participants) | 197
Participants
  ADA negative or ADA positive with no boost | 170
  Induced or Boosted | 27

43. Secondary Outcome: Pharmacokinetic Parameters: Cmax After First Brolucizumab 6 mg Dose in a Subset of Subjects
Description: The maximum (peak) observed serum drug concentration after single dose administration (mass x volume-1)
Time Frame: Day 1, Day 2, Day 8, Day 15, Day 22, and Day 29
Population: Safety Analysis Set - for a subset of participants with a valid measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 13 | 0
ng/mL | 39.7 (121.0) |

44. Secondary Outcome: Pharmacokinetic Parameters: Tmax After First Brolucizumab 6 mg Dose in a Subset of Subjects
Description: The time to reach maximum (peak) serum drug concentration after single dose administration (time).
  Actual sampling times were taken into consideration for the pharmacokinetic (PK) analysis.
Time Frame: Day 1, Day 2, Day 8, Day 15, Day 22, and Day 29
Population: Safety Analysis Set - for a subset of participants with a valid measurement
Measure: Median (Full Range); unit: hour
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 13 | 0
hour | 5.25 [5.03 to 20.3] |

45. Secondary Outcome: Pharmacokinetic Parameters: AUClast After First Brolucizumab 6 mg Dose in a Subset of Subjects
Description: The AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1)
Time Frame: Day 1, Day 2, Day 8, Day 15, Day 22, and Day 29
Population: Safety Analysis Set - for a subset of treated participants with a valid measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 13 | 0
h*ng/mL | 2690 (74.4) |

46. Secondary Outcome: Pharmacokinetic Parameters: AUCinf After First Brolucizumab 6 mg Dose in a Subset of Subjects
Description: The AUC from time zero to infinity (mass x time x volume-1)
Time Frame: Day 1, Day 2, Day 8, Day 15, Day 22, and Day 29
Population: Safety Analysis Set - for a subset of treated participants with a valid measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 11 | 0
h*ng/mL | 3100 (73.4) |

47. Secondary Outcome: Pharmacokinetic Parameters: T1/2 After First Brolucizumab 6 mg Dose in a Subset of Subjects
Description: The elimination half-life associated with the terminal slope (lz) of a semi logarithmic concentration time curve (time).
Time Frame: Day 1, Day 2, Day 8, Day 15, Day 22, and Day 29
Population: Safety Analysis Set - for a subset of treated participants with a valid measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 11 | 0
hours | 110 (37.9) |

48. Secondary Outcome: Pharmacokinetic Parameters: CL/F After First Brolucizumab 6 mg Dose in a Subset of Subjects
Description: Apparent total body clearance of siremadlin from serum (CL/F)
Time Frame: Day 1, Day 2, Day 8, Day 15, Day 22, and Day 29
Population: Safety Analysis Set - for a subset of treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 11 | 0
Liters/hour | 1.93 (73.4) |

49. Secondary Outcome: Pharmacokinetic Parameters: Vz/F After First Brolucizumab 6 mg Dose in a Subset of Subjects
Description: Apparent volume of distribution during terminal elimination phase (Vz/F)
Time Frame: Day 1, Day 2, Day 8, Day 15, Day 22, and Day 29
Population: Safety Analysis Set - for a subset of treated participants with a valid measurement
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 11 | 0
L | 307 (48.6) |

50. Secondary Outcome: Most Common Ocular Adverse Events (Greater Than or Equal to 2% in Any Treatment Arm) by Preferred Term for the Study Eye
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  Treatment-emergent AEs are presented, which are AEs that developed on or after first study treatment administration, or any event previously present that worsened following exposure to the study treatment.
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum timeframe of approximately 48 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  Number of participants with at least one AE | 58 | 48
  Intraocular pressure increased | 10 | 6
  Conjunctival haemorrhage | 7 | 3
  Visual acuity reduced | 7 | 2
  Retinal haemorrhage | 6 | 4
  Uveitis | 6 | 0
  Conjunctivitis | 5 | 4
  Dry eye | 5 | 3
  Cataract | 4 | 8
  Meibomian gland dysfunction | 4 | 7
  Xerophthalmia | 4 | 2

51. Secondary Outcome: Non-ocular Adverse Events (Greater Than or Equal to 2% in Any Treatment Arm)
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  Treatment-emergent AEs are counted, which are AEs that developed on or after first study treatment administration, or any event previously present that worsened following exposure to the study treatment.
Time Frame: as for outcome 50
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants | 97 | 113

52. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum timeframe of approximately 48 weeks.
  Post-treatment deaths are reported 30 days after last treatment to 72 days post treatment (Day 185).
Time Frame: Deaths are reported from first dose of study treatment until approximately Day 185.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 199 | 198
Participants
  On-treatment Deaths | 0 | 0
  Post-treatment Deaths | 0 | 1
  Total Deaths | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum timeframe of approximately 48 weeks. Deaths are reported from first dose of study treatment until approximately Day 185.
Groups:
- Brolucizumab 6mg: 3 monthly intravitreal injections of brolucizumab 6 mg in the loading treatment period (q4w regimen) up to Week 8 followed by injections every 12 weeks (q12w regimen) or 8 weeks (q8w) up to Week 40 or Week 44, depending on disease activity status.
- Aflibercept 2mg: 3 monthly intravitreal injections of aflibercept 2 mg in the loading treatment period (q4w regimen) up to Week 8 followed by injections every 8 weeks (q8w) up to Week 40.
- Overall: Overall
Arm/Group | Brolucizumab 6mg | Aflibercept 2mg | Overall
All-Cause Mortality (participants affected / at risk) | 0/199 | 1/198 | 1/397
Serious Adverse Events (participants affected / at risk) | 23/199 | 24/198 | 47/397
Other Adverse Events (participants affected / at risk) | 94/199 | 90/198 | 184/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=199) | Aflibercept 2mg (N=198) | Overall (N=397)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 1
Cataract - Fellow eye (Eye disorders) | 1 | 0 | 1
Cataract - Study eye (Eye disorders) | 1 | 0 | 1
Iridodialysis - Study eye (Eye disorders) | 1 | 0 | 1
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 1 | 0 | 1
Vitreous haemorrhage - Fellow eye (Eye disorders) | 0 | 1 | 1
Vitreous haemorrhage - Study eye (Eye disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 2 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 2
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Corneal laceration - Study eye (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Malignant mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 2
Cerebral infarction (Nervous system disorders) | 2 | 2 | 4
Lacunar infarction (Nervous system disorders) | 2 | 1 | 3
Thalamic infarction (Nervous system disorders) | 0 | 1 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 1 | 2
Device breakage (Product Issues) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=199) | Aflibercept 2mg (N=198) | Overall (N=397)
Arteriosclerosis coronary artery (Cardiac disorders) | 5 | 1 | 6
Thyroid mass (Endocrine disorders) | 4 | 0 | 4
Cataract - Fellow eye (Eye disorders) | 2 | 5 | 7
Cataract - Study eye (Eye disorders) | 3 | 8 | 11
Conjunctival haemorrhage - Study eye (Eye disorders) | 7 | 3 | 10
Dry eye - Fellow eye (Eye disorders) | 5 | 4 | 9
Dry eye - Study eye (Eye disorders) | 5 | 3 | 8
Meibomian gland dysfunction - Fellow eye (Eye disorders) | 4 | 6 | 10
Meibomian gland dysfunction - Study eye (Eye disorders) | 4 | 7 | 11
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 1 | 7 | 8
Retinal haemorrhage - Study eye (Eye disorders) | 6 | 4 | 10
Uveitis - Study eye (Eye disorders) | 6 | 0 | 6
Visual acuity reduced - Study eye (Eye disorders) | 7 | 2 | 9
Xerophthalmia - Fellow eye (Eye disorders) | 4 | 2 | 6
Xerophthalmia - Study eye (Eye disorders) | 4 | 2 | 6
Pyrexia (General disorders) | 8 | 7 | 15
COVID-19 (Infections and infestations) | 22 | 26 | 48
Conjunctivitis - Study eye (Infections and infestations) | 5 | 4 | 9
Pneumonia (Infections and infestations) | 5 | 4 | 9
Upper respiratory tract infection (Infections and infestations) | 15 | 14 | 29
Urinary tract infection (Infections and infestations) | 0 | 5 | 5
Blood urea nitrogen/creatinine ratio increased (Investigations) | 4 | 3 | 7
Intraocular pressure increased - Fellow eye (Investigations) | 3 | 5 | 8
Intraocular pressure increased - Study eye (Investigations) | 10 | 6 | 16
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 5 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 6
Renal cyst (Renal and urinary disorders) | 4 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 11
Aortic arteriosclerosis (Vascular disorders) | 4 | 1 | 5
Hypertension (Vascular disorders) | 6 | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT04047472/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT04047472/SAP_001.pdf